CLINICAL TRIAL: NCT02191137
Title: A Phase IV, Prospective, Single-Arm, Open-Label Study to Measure Outcomes in Patients With Pulmonary Arterial Hypertension Not on Active Treatment
Brief Title: Measuring Outcomes In Patients With Pulmonary Arterial Hypertension Not on Active Treatment (MOTION)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17407
Record Dates: First submitted 2014-06-27; First posted 2014-07-16 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-09

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary Hypertension,Riociguat,Living with Pulmonary Hypertension Questionnaire
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Riociguat 0.5mg to 2.5 mg (Experimental): Single arm, open label
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — Participants received therapy with riociguat during a 10-week titration phase. The starting dose for riociguat for all patients was 0.5 milligram (mg) three times a day (TID). The dose of riociguat was increased every 2 weeks in 0.5 mg increments to 1.0, 1.5, 2.0, and 2.5 mg until patients reached their individual optimal dose based on their systolic blood pressure and well-being. After reaching their optimal dose, patients then entered a maintenance phase and remained on this dose for an additional 14 weeks. End of treatment was reached at Visit 10 after 24 weeks of treatment with riociguat.

SUMMARY:
The MOTION study was a prospective, Phase IV study for patients with Pulmonary Arterial Hypertension (PAH). The study was designed to further explore patient-reported outcomes in PAH subjects who were not on active treatment and living in the United States. In addition, the study explored the use of new telemetric technology (Accelerator band) to evaluate if this technology correlates with improvements in 6 Minute Walking Distance 6MWD in patients with PAH.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 18 to 80 years of age at Visit 0
* Women of childbearing potential must have a negative pre-treatment pregnancy test, negative monthly pregnancy test, and must use reliable methods of contraception according to the Risk Evaluation Mitigation Strategies (REMS) guidance
* Symptomatic pulmonary arterial hypertension, World Health Organization Group 1 with a pulmonary vascular resistance (PVR) >300 dyn*sec*cm-5, mean pulmonary artery pressure (PAP mean) ≥25 mmHg, and pulmonary capillary wedge pressure (PCWP) ≤15 mmHg as assessed by right heart catheterization within 6 months prior to Screening (Visit 0)
* PAH of the following types:

Idiopathic (IPAH) Familial (FPAH)

Associated with PAH (APAH) due to:

Connective tissue disease Congenital heart disease, but only if patient underwent surgical repair more than one year before enrollment Anorexigen or amphetamine use Portal hypertension with liver cirrhosis

* Not treated with PAH-specific pulmonary medications within 14 days of Screening (Visit 0)
* 6MWD between 150 meters and 450 meters

Exclusion Criteria:

* Patients who are pregnant
* Patients currently on nitrate and/or nitric oxide (NO) donor therapy; patients currently taking phosphodiesterase 5 (PDE5) inhibitors (such as sildenafil, tadalafil, vardenafil) and non-specific PDE inhibitors (theophylline, dipyridamole)
* Non-WHO group 1 Pulmonary Hypertension
* Severe restrictive lung disease
* History of uncontrolled high blood pressure or hypotension
* A medical disorder, condition, or history that in the opinion of the Investigator would impair their ability to participate or complete this study
* Active state of hemoptysis or pulmonary hemorrhage, including those events managed by bronchial artery embolization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2016-07-16 (Actual); Study Completion 2016-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (55):
- United States (54):
  - Tucson, Arizona
  - La Jolla, California
  - Moreno Valley, California
  - Pomona, California
  - Sacramento, California
  - San Juan Capistrano, California
  - Santa Barbara, California
  - Aurora, Colorado
  - Hartford, Connecticut
  - Celebration, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Orlando, Florida
  - Weston, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Austell, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Fort Wayne, Indiana
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - North Dartmouth, Massachusetts
  - Detroit, Michigan
  - Troy, Michigan
  - Pascagoula, Mississippi
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Newark, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Brooklyn, New York
  - Liverpool, New York
  - Mineola, New York
  - New Hyde Park, New York
  - Stony Brook, New York
  - Syracuse, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Sioux Falls, South Dakota
  - El Paso, Texas
  - Houston, Texas
  - Temple, Texas
  - Milwaukee, Wisconsin
- Guaynabo, Puerto Rico

REFERENCES:
- [Derived] Mathai SC, Minai O, Sullivan SD, Lerner D, Levine D. Rationale and study design of MOTION: A phase 4, prospective, single-arm, open-label study to measure outcomes in patients with pulmonary arterial hypertension not on active treatment. Respir Med. 2017 Jan;122 Suppl 1:S23-S27. doi: 10.1016/j.rmed.2016.11.002. Epub 2016 Nov 2. PMID 27890471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 97 patients signed informed consent; 22 patients did not complete screening (20 patients were screen failures and 2 patients withdrew from the study). Of 75 patients who received therapy with riociguat, 65 patients completed study treatment and entered follow-up, and 60 patients completed the study.
Period: Treatment
Arm/Group | Riociguat (Adempas, BAY63-2521)
Started | 75
Completed | 65
Not Completed | 10
Not completed — Death | 4
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 2
Not completed — Other | 1
Period: Follow-up
Arm/Group | Riociguat (Adempas, BAY63-2521)
Started | 65
Completed | 60
Not Completed | 5
Not completed — Lost to Follow-up | 2
Not completed — Ongoing/unknown | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 9
Living with Pulmonary Hypertension (LPH) [Mean (Standard Deviation); unit: Scores] — The LPH derived from the Minnesota Living with Heart Failure questionnaire comprises 21 items, responded to on a 6-point Likert scale ranging from 0 'No' to 5 'Very much'. A total score ranging from 0 to 105 is calculated by summing the responses to all 21 questions. A physical dimension score (range 0-40, 8 items) and an emotional dimension score (range 0-25, 5 items) can also be calculated. For all LPH scores, a higher score indicates that patients are more affected by their medical condition.
  Scores
    Total score | 46.03 (24.57)
    Physical dimension score | 22.83 (10.70)
    Emotional dimension score | 10.20 (7.80)
Short Form-12 Health Survey (SF-12) questionnaire [Mean (Standard Deviation); unit: Scores]
  Physical component summary | 36.660 (8.577)
  Mental component summary | 47.453 (9.213)
WHO functional class [Number; unit: Percentage of participants]
  I | 9.3
  II | 30.7
  III | 58.7
  IV | 1.3
Modified Borg Dyspnea Scale [Mean (Standard Deviation); unit: Scores] | 4.47 (2.74)
Six-minute walk distance (6MWD) [Mean (Standard Deviation); unit: Meters] | 310.259 (89.578)
Work Limitations Questionnaire (WLQ) [Mean (Standard Deviation); unit: Percentage] — The Work Limitations Questionnaire (WLQ) is an 8-item questionnaire that measures the degree to which employed individuals are experiencing limitations on-the-job due to their health problems, and health-related productivity loss (Presenteeism). The WLQ's terms are aggregated into four scales (i.e. Time Management, Physical demands, Mental-interpersonal demands, Output demands). Scale score range from 0 (limited none of the time) to 100 (limited all of the time) and represent the reported amount of time in the prior two weeks respondents were limited on-the-job.
  Percentage
    Time management scale | 36.42 (30.82)
    Physical demands scale | 33.47 (28.25)
    Mental-interpersonal demands scale | 28.66 (25.22)
    Output demands scale | 36.52 (31.51)
WLQ: Percentage of Productivity loss [Mean (Standard Deviation); unit: Percentage] — The WLQ is an 8-item questionnaire that measures the degree to which employed individuals are experiencing limitations on-the-job due to their health problems, and health-related productivity loss (Presenteeism). The WLQ's terms are aggregated into four scales (i.e. Time Management, Physical demands, Mental-interpersonal demands, Output demands). Using an algorithm, WLQ scale scores can be converted into an estimate of productivity loss.
  Percentage | 8.85 (6.62)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in the Living With Pulmonary Hypertension (LPH) Questionnaire Total Score
Description: The Living with Pulmonary Hypertension (LPH) questionnaire with Heart Failure questionnaire comprises 21 items, responded to on a 6-point Likert scale ranging from 0 'No' to 5 'Very much'. A total score ranging from 0 (best) to 105 (worst) is calculated by summing the responses to all 21 questions.
Time Frame: Baseline to Week 24
Population: The ITT analysis set was synonymous with the Safety analysis set definition which included all patients who received at least 1 dose of test drug. 66 patients were evaluable for LPH total score at Week 24.
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 66
Scores | -10.99 (22.51)

2. Secondary Outcome: Change From Baseline to Weeks 4 and 16 in the LPH Total Score
Description: The Living with Pulmonary Hypertension (LPH) questionnaire with Heart Failure questionnaire comprises 21 items, responded to on a 6-point Likert scale ranging from 0 'No' to 5 'Very much'. A total score ranging from 0 (best) to 105 (worst) is calculated by summing the responses to all 21 questions. In the below table, "N" signifies subjects who were evaluable for the specific parameter at that timepoint.
Time Frame: Baseline to Week 4 and Week 16
Population: The ITT analysis set was synonymous with the Safety analysis set definition which included all patients who received at least 1 dose of test drug. 72 patients were evaluable for LPH total score at Week 4.
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 72
Scores
  Week 4 (N=72) | -7.65 (18.30)
  Week 16 (N=68) | -6.98 (20.85)

3. Secondary Outcome: Change From Week 16 to Week 24 in the LPH Total Score (Completers Analysis Set Only)
Description: as for outcome 1
Time Frame: Week 16 to Week 24
Population: The Completers analysis set included patients valid for Safety/ITT analysis sets who had an LPH score at baseline (Visit 1), Week 4, Week 16, and Week 24. 58 patients in Completer analysis set were evaluable for LPH total score at Week 24.
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 58
Scores | -1.66 (15.13)

4. Secondary Outcome: Change From Baseline to Weeks 4, 16, and 24 in the LPH Physical Dimension Score
Description: The LPH derived from the Minnesota Living with Heart Failure questionnaire comprises 21 items, responded to on a 6-point Likert scale ranging from 0 'No' to 5 'Very much'. A total score ranging from 0 to 105 is calculated by summing the responses to all 21 questions. A physical dimension score (range 0-40, 8 items) and an emotional dimension score (range 0-25, 5 items) can also be calculated. For all LPH scores, a higher score indicates that patients are more affected by their medical condition. In the below table, "N" signifies subjects who were evaluable for the specific parameter at that timepoint.
Time Frame: Baseline to Weeks 4, 16, and 24
Population: The ITT analysis set was synonymous with the Safety analysis set definition which included all patients who received at least 1 dose of test drug. 75 patients were evaluable for LPH physical dimension score at week 16 or before.
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 75
Scores
  Week 4 (N=72) | -3.77 (8.25)
  Week 16 or Last Before (N=75) | -3.97 (9.94)
  Week 24 (N=65) | -6.10 (9.38)

5. Secondary Outcome: Change From Week 16 to Week 24 in the LPH Physical Dimension Score (Completers Analysis Set Only)
Description: The LPH derived from the Minnesota Living with Heart Failure questionnaire comprises 21 items, responded to on a 6-point Likert scale ranging from 0 'No' to 5 'Very much'. A total score ranging from 0 to 105 is calculated by summing the responses to all 21 questions. A physical dimension score (range 0-40, 8 items) and an emotional dimension score (range 0-25, 5 items) can also be calculated. For all LPH scores, a higher score indicates that patients are more affected by their medical condition.
Time Frame: Week 16 to Week 24
Population: The Completers analysis set included patients valid for Safety/ITT analysis sets who had an LPH score at baseline (Visit 1), Week 4, Week 16, and Week 24. 57 patients in Completer analysis set were evaluable for LPH physical dimension score at Week 24.
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 57
Scores | -0.86 (7.20)

6. Secondary Outcome: Change From Baseline to Weeks 4, 16, and 24 in the LPH Emotional Dimension Score
Description: as for outcome 4
Time Frame: Baseline to Week 4, Week 16 and Week 24
Population: The ITT analysis set was synonymous with the Safety analysis set definition which included all patients who received at least 1 dose of test drug. 75 patients were evaluable for LPH emotional dimension score at week 16 or before.
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 75
Scores
  Week 4 (N=72) | -2.22 (5.70)
  Week 16 or Last Before (N=75) | -1.44 (7.32)
  Week 24 (N=66) | -2.33 (6.90)

7. Secondary Outcome: Change From Week 16 to Week 24 in the LPH Emotional Dimension Score (Completers Analysis Set Only)
Description: as for outcome 5
Time Frame: Week 16 to Week 24
Population: The Completers analysis set included patients valid for Safety/ITT analysis sets who had an LPH score at baseline (Visit 1), Week 4, Week 16, and Week 24. 58 patients in Completer analysis set were evaluable for LPH emotional dimension score at Week 24.
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 58
Scores | -0.11 (5.50)

8. Secondary Outcome: Percentage of Patients With a Minimal Clinically Significant Important Difference (MCID) From Baseline in LPH Total Score at Weeks 4, 16, and 24
Description: For LPH total score, the MCID was an 11-point decrease from baseline. In the below table, "N" signifies subjects who were evaluable for the specific parameter at that timepoint.
Time Frame: Baseline to Week 4, Week 16 and Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 72
Percentage of participants
  Week 4 (N=72) | 38.9 [0.34 to 0.58]
  Week 16 (N=68) | 45.6 [0.39 to 0.64]
  Week 24 (N=66) | 47.0 [0.47 to 0.72]

9. Secondary Outcome: Percentage of Patients With an MCID From Baseline in LPH Physical Dimension Score at Weeks 4, 16, and 24
Description: For the physical and emotional dimension scores, the MCID was a 4-point decrease. In the below table, "N" signifies subjects who were evaluable for the specific parameter at that timepoint.
Time Frame: Baseline to Week 4, Week 16 and Week 24
Population: The ITT analysis set was synonymous with the Safety analysis set definition which included all patients who received at least 1 dose of test drug. 72 patients were evaluable for LPH physical dimension score at week 4.
Measure: Number; unit: Percentage of Participants
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 72
Percentage of Participants
  Week 4 (N=72) | 45.8
  Week 16 (N=68) | 51.5
  Week 24 (N=65) | 60.0

10. Secondary Outcome: Percentage of Patients With an MCID From Baseline in LPH Emotional Dimension Score at Weeks 4, 16, and 24
Description: as for outcome 9
Time Frame: Baseline to Week 4, Week 16 and Week 24
Population: The ITT analysis set was synonymous with the Safety analysis set definition which included all patients who received at least 1 dose of test drug. 72 patients were evaluable for LPH emotional dimension score at week 4.
Measure: Number; unit: Percentage of Participants
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 72
Percentage of Participants
  Week 4 (N=72) | 31.9
  Week 16 (N=68) | 39.7
  Week 24 (N=66) | 33.3

11. Secondary Outcome: Percentage of Patients With an MCID From Week 16 in LPH Total Score at Week 24 (Completers Analysis Set Only)
Description: For LPH total score, the MCID was an 11-point decrease.
Time Frame: Week 16 to Week 24
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 58
Percentage of Participants | 24.1

12. Secondary Outcome: Percentage of Patients With an MCID From Week 16 in Physical Dimension Score at Week 24 (Completers Analysis Set Only)
Description: For the physical and emotional dimension scores, the MCID was a 4-point decrease.
Time Frame: Week 16 to Week 24
Population: The Completers analysis set included patients valid for Safety/ITT analysis sets who had an LPH score at baseline (Visit 1), Week 4, Week 16, and Week 24. 57 patients were evaluable for LPH physical dimension score at week 24.
Measure: Number; unit: Percentage of Participants
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 57
Percentage of Participants | 29.8

13. Secondary Outcome: Percentage of Patients With an MCID From Week 16 in Emotional Dimension Score at Week 24 (Completers Analysis Set Only)
Description: For the physical and emotional dimension scores, the MCID was a 4-point decrease.
Time Frame: Week 16 to Week 24
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 58
Percentage of Participants | 17.2

14. Secondary Outcome: Change From Baseline to Weeks 4, 16, and 24 in the WLQ Time Management, Physical Demands, Mental-Interpersonal Demands and Output Demands Scores
Description: The Work Limitations Questionnaire (WLQ) is an 8-item questionnaire that measures the degree to which employed individuals are experiencing limitations on-the-job due to their health problems, and health-related productivity loss (Presenteeism). The WLQ's terms are aggregated into four scales (i.e. Time Management, Physical demands, Mental-interpersonal demands, Output demands). Scale score range from 0 (limited none of the time) to 100 (limited all of the time) and represent the reported amount of time in the prior two weeks respondents were limited on-the-job. In the below table, "N" signifies subjects who were evaluable for the specific parameter at that timepoint.
Time Frame: Baseline to Week 4, Week 16 and Week 24
Population: The ITT analysis set was synonymous with the Safety analysis set definition which included all patients who received at least 1 dose of test drug. 52 patients were evaluable for WLQ at week 4.
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 52
Scores
  Week 4 Time management score, N=45 | 4.17 (25.28)
  Week 4 Physical demands score, N=52 | 0.96 (25.35)
  Week 4 Mental-interpersonal demands score, N=48 | -8.59 (25.29)
  Week 4 Output demands score, N=40 | -6.88 (27.00)
  Week 16 Time management score, N=45 | 0.56 (26.24)
  Week 16 Physical demands score, N=49 | 7.40 (26.26)
  Week 16 Mental-interpersonal demands score, N=46 | -6.52 (24.82)
  Week 16 Output demands score, N=40 | 2.81 (25.71)
  Week 24 Time management score, N=42 | -2.68 (26.41)
  Week 24 Physical demands score, N=43 | 2.33 (21.17)
  Week 24 Mental-interpersonal demands score, N=41 | -2.13 (25.91)
  Week 24 Output demands score, N=34 | -2.57 (25.71)

15. Secondary Outcome: Change From Baseline to Weeks 4, 16, and 24 in the WLQ Percentage of Productivity Loss
Description: The WLQ is an 8-item questionnaire that measures the degree to which employed individuals are experiencing limitations on-the-job due to their health problems, and health-related productivity loss (Presenteeism). The WLQ's terms are aggregated into four scales (i.e. Time Management, Physical demands, Mental-interpersonal demands, Output demands). Using an algorithm, WLQ scale scores can be converted into an estimate of productivity loss. In the below table, "N" signifies subjects who were evaluable for the specific parameter at that timepoint.
Time Frame: Baseline to Week 4, Week 16 and Week 24
Population: The ITT analysis set was synonymous with the Safety analysis set definition which included all patients who received at least 1 dose of test drug. 37 patients were evaluable for WLQ percentage of productivity loss at week 4.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 52
Percentage
  Week 4 Productivity loss (%), N=37 | -1.07 (4.68)
  Week 16 Productivity loss (%), N=30 | 0.54 (4.85)
  Week 24 Productivity loss (%), N=27 | -0.53 (5.82)

16. Secondary Outcome: Change From Week 16 to Week 24 in the WLQ Time Management, Physical Demands, Mental-Interpersonal Demands, and Output Demands Scores (Completers Analysis Set Only)
Description: The Work Limitations Questionnaire (WLQ) is an 8-item questionnaire that measures the degree to which employed individuals are experiencing limitations on-the-job due to their health problems, and health-related productivity loss (Presenteeism). The WLQ's terms are aggregated into four scales (i.e. Time Management, Physical demands, Mental-interpersonal demands, Output demands). Scale score range from 0 (limited none of the time) to 100 (limited all of the time) and represent the reported amount of time in the prior two weeks respondents were limited on-the-job.
Time Frame: Week 16 to Week 24
Population: The Completers analysis set included patients valid for Safety/ITT analysis sets who had an LPH score at baseline (Visit 1), Week 4, Week 16, and Week 24. 40 patients in Completer analysis set were evaluable for WLQ at Week 24.
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 40
Scores
  Time management score, N=39 | -0.32 (25.73)
  Physical demands score, N=40 | -1.56 (24.22)
  Mental-interpersonal demands score, N=38 | 5.92 (19.87)
  Output demands score, N=34 | -4.78 (24.43)

17. Secondary Outcome: Change From Week 16 to Week 24 in the WLQ Percentage of Productivity Loss (Completers Analysis Set Only)
Description: The WLQ is an 8-item questionnaire that measures the degree to which employed individuals are experiencing limitations on-the-job due to their health problems, and health-related productivity loss (Presenteeism). The WLQ's terms are aggregated into four scales (i.e. Time Management, Physical demands, Mental-interpersonal demands, Output demands). Using an algorithm, WLQ scale scores can be converted into an estimate of productivity loss.
Time Frame: Week 16 to Week 24
Population: The Completers analysis set included patients valid for Safety/ITT analysis sets who had an LPH score at baseline (Visit 1), Week 4, Week 16, and Week 24. 40 patients in Completer analysis set were evaluable for WLQ percentage of productivity loss at week 24.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 40
Percentage | 0.19 (4.17)

18. Secondary Outcome: Change From Baseline to Weeks 4, 16, and 24 in the Short Form-12 Health Survey (SF-12) Physical Component Summary (PCS) Score and Mental Component Summary (MCS) Score
Description: SF-12v2® Health Survey is a 12-item questionnaire to measure functional health and well-being from the patient's point of view. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. In the below table, "N" signifies subjects who were evaluable for the specific parameter at that timepoint.
Time Frame: Baseline to Week 4, Week 16 and Week 24
Population: The ITT analysis set was synonymous with the Safety analysis set definition which included all patients who received at least 1 dose of test drug. 73 patients were evaluable for PCS and MCS at Week 4.
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 73
Scores
  PCS Week 4 (N=73) | 1.009 (6.474)
  PCS Week 16 (N=69) | 0.036 (7.059)
  PCS Week 24 (N=67) | 1.230 (8.401)
  MCS Week 4 (N=73) | 1.955 (9.262)
  MCS Week 16 (N=69) | 1.869 (7.605)
  MCS Week 24 (N=67) | 2.883 (10.073)

19. Secondary Outcome: Change From Week 16 to Week 24 in the SF-12 PCS Score and MCS Score (Completers Analysis Set Only)
Description: SF-12v2® Health Survey is a 12-item questionnaire to measure functional health and well-being from the patient's point of view. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Week 16 to Week 24
Population: The Completers analysis set included patients valid for Safety/ITT analysis sets who had an LPH score at baseline (Visit 1), Week 4, Week 16, and Week 24. 58 patients in Completer analysis set were evaluable for PCS and MCS at Week 24.
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 58
Scores
  PCS | 1.383 (6.810)
  MCS | 0.437 (8.378)

20. Secondary Outcome: Change From Baseline to Weeks 4, 16, and 24 in the WHO Functional Class
Description: Functional class was determined by the WHO classification:
  I: Patients with PH (pulmonary hypertension) but without resulting limitation of physical activity. Ordinary physical activity does not cause undue dyspnea or fatigue, chest pain, or near syncope.
  II: Patients with PH resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity causes undue dyspnea or fatigue, chest pain, or near syncope.
  III: Patients with PH resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes undue dyspnea or fatigue, chest pain, or near syncope.
  IV: Patients with PH with inability to carry out any physical activity without symptoms. These patients manifest signs of right-heart failure. Dyspnea and/or fatigue may even be present at rest. Discomfort is increased by any physical activity.
  In the below table, "N" signifies subjects who were evaluable for the specific parameter at that timepoint.
Time Frame: Baseline to Week 4, Week 16 and Week 24
Population: The ITT analysis set was synonymous with the Safety analysis set definition which included all patients who received at least 1 dose of test drug. 75 patients were evaluable for WHO Function Class at Week 16 or Last Before.
Measure: Number; unit: Percentage of participants
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 75
Percentage of participants
  Week 4 (-1 Change in WHO Class), N=72 | 9.7
  Week 4 (0 Change in WHO Class), N=72 | 87.5
  Week 4 (+1 Change in WHO Class), N=72 | 2.8
  Week 4 (+2 Change in WHO Class), N=72 | 0
  Week 16 or LastBefore (-1 Change in WHOClass),N=75 | 18.7
  Week 16 or LastBefore (0 Change in WHOClass),N=75 | 66.7
  Week 16 or LastBefore (+1 Change in WHOClass),N=75 | 12.0
  Week 16 or LastBefore (+2 Change in WHOClass),N=75 | 2.7
  Week 24 (-1 Change in WHO Class), N=67 | 28.4
  Week 24 (0 Change in WHO Class), N=67 | 64.2
  Week 24 (+1 Change in WHO Class), N=67 | 6.0
  Week 24 (+2 Change in WHO Class), N=67 | 1.5

21. Secondary Outcome: Change From Week 16 to Week 24 in the WHO Functional Class (Completers Analysis Set Only)
Description: Functional class was determined by the WHO classification:
  I: Patients with PH (pulmonary hypertension) but without resulting limitation of physical activity. Ordinary physical activity does not cause undue dyspnea or fatigue, chest pain, or near syncope.
  II: Patients with PH resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity causes undue dyspnea or fatigue, chest pain, or near syncope.
  III: Patients with PH resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes undue dyspnea or fatigue, chest pain, or near syncope.
  IV: Patients with PH with inability to carry out any physical activity without symptoms. These patients manifest signs of right-heart failure. Dyspnea and/or fatigue may even be present at rest. Discomfort is increased by any physical activity.
Time Frame: Week 16 to Week 24
Population: The Completers analysis set included patients valid for Safety/ITT analysis sets who had an LPH score at baseline (Visit 1), Week 4, Week 16, and Week 24. 57 patients in Completer analysis set were evaluable for WHO Function Class at Week 24.
Measure: Number; unit: Percentage of participants
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 57
Percentage of participants
  -2 Change in WHO Class | 1.8
  -1 Change in WHO Class | 15.8
  0 Change in WHO Class | 70.2
  +1 Change in WHO Class | 10.5
  +2 Change in WHO Class | 1.8

22. Secondary Outcome: Change From Baseline to Weeks 16 and 24 in the Modified Borg Dyspnea Scale
Description: The Modified Borg Dyspnea Scale assessed the intensity of the patient's dyspnea from 0 (best) to 10 (worst). In the below table, "N" signifies subjects who were evaluable for the specific parameter at that timepoint.
Time Frame: Week 16 to Week 24
Population: The ITT analysis set was synonymous with the Safety analysis set definition which included all patients who received at least 1 dose of test drug. 58 patients were evaluable for Modified Borg Dyspnea Scale at week 24.
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 58
Scores
  Week 16 (N=57) | -0.70 (3.23)
  Week 24 (N=58) | -0.91 (3.44)

23. Secondary Outcome: Change From Week 16 to Week 24 in the Modified Borg Dyspnea Scale (Completers Analysis Set Only)
Description: The Modified Borg Dyspnea Scale assessed the intensity of the patient's dyspnea from 0 (best) to 10 (worst).
Time Frame: Week 16 to Week 24
Population: The Completers analysis set included patients valid for Safety/ITT analysis sets who had an LPH score at baseline (Visit 1), Week 4, Week 16, and Week 24. 57 patients in Completer analysis set were evaluable for Modified Borg Dyspnea Scale at Week 24.
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 57
Scores | -0.19 (3.75)

24. Secondary Outcome: Change From Baseline to Weeks 16 and 24 in the 6MWD
Description: Six-minute walk distance (6MWD) was conducted to test the physical limitations of the patient by assessing the patient's exercise capacity. The distance walked by the patient in 6 minutes was measured. In the below table, "N" signifies subjects who were evaluable for the specific parameter at that timepoint.
Time Frame: Week 16 to Week 24
Population: The ITT analysis set was synonymous with the Safety analysis set definition which included all patients who received at least 1 dose of test drug. 67 patients were evaluable for 6MWD at week 24.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 67
Meters
  Week 16 (N=66) | 2.362 (75.506)
  Week 24 (N=67) | -2.921 (59.247)

25. Secondary Outcome: Change From Week 16 to Week 24 in the 6MWD (Completers Analysis Set Only)
Description: Six-minute walk distance (6MWD) was conducted to test the physical limitations of the patient by assessing the patient's exercise capacity. The distance walked by the patient in 6 minutes was measured.
Time Frame: Week 16 to Week 24
Population: The Completers analysis set included patients valid for Safety/ITT analysis sets who had an LPH score at baseline (Visit 1), Week 4, Week 16, and Week 24. 57 patients in Completer analysis set were evaluable for 6MWD at week 24.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 57
Meters | -7.932 (71.542)

ADVERSE EVENTS:
Time Frame: From the first dose of test drug up to 2 days after the last dose.
Arm/Group | Riociguat (Adempas, BAY63-2521)
Serious Adverse Events (participants affected / at risk) | 21/75
Other Adverse Events (participants affected / at risk) | 61/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riociguat (Adempas, BAY63-2521) (N=75)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 3 (4)
Sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riociguat (Adempas, BAY63-2521) (N=75)
Palpitations (Cardiac disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 14 (18)
Dyspepsia (Gastrointestinal disorders) | 15 (24)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 16 (18)
Vomiting (Gastrointestinal disorders) | 9 (10)
Chest pain (General disorders) | 8 (8)
Fatigue (General disorders) | 10 (10)
Oedema peripheral (General disorders) | 9 (10)
Peripheral swelling (General disorders) | 4 (4)
Bronchitis (Infections and infestations) | 4 (4)
Influenza (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 9 (9)
Pneumonia (Infections and infestations) | 4 (4)
Sinusitis (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Dizziness (Nervous system disorders) | 17 (20)
Headache (Nervous system disorders) | 13 (15)
Insomnia (Psychiatric disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypotension (Vascular disorders) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less